CLINICAL TRIAL: NCT06315413
Title: Evaluation of Socket Seal Using Flowable Composite Above Xenograft Compared to Dense Polytetrafluoroethylene (d-PTFE) Membrane in Ridge Preservation Procedures: a Randomized Controlled Clinical Trial
Brief Title: Composite Plug Vs D-PTFE Membrane in Socket Preservation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Youssef Emad Zaghloul Meshreky, Assistant lecturer of Periodontology, Newgiza University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Composite plug vs d-PTFE
Record Dates: First submitted 2024-03-10; First posted 2024-03-18 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-08

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Composite plug (Experimental): Tooth extraction will be done a-traumatically followed by socket curettage and cleaning followed by xenograft filling for the socket and coverage with injected flowable composite plug which will then be stabilized using 5.0 polypropylene suture material with a figure of eight suture.
  Interventions: Procedure: Socket preservation using xenograft and composite plug
- Exposed d-PTFE (Active Comparator): Tooth extraction will be done a-traumatically followed by socket curettage and cleaning followed by xenograft filling for the socket and coverage with d-PTFE membrane which will be left exposed intentionally and secured using 5.0 polypropylene suture material with a figure of eight suture.
  Interventions: Procedure: Socket preservation using xenograft and intentionally exposed d-PTFE

INTERVENTIONS:
Procedure: Socket preservation using xenograft and composite plug — Extraction of hopeless teeth will be followed by grafting the socket with xenograft and coverage with injected flowable composite plug which will then be stabilized using 5.0 polypropylene suture material with a figure of eight suture.
  Arms: Composite plug
Procedure: Socket preservation using xenograft and intentionally exposed d-PTFE — Extraction of hopeless teeth will be followed by grafting the socket with xenograft and coverage with d-PTFE membrane which will the be left exposed intentionally. This will be followed by securing the membrane using 5.0 polypropylene suture material with a figure of eight suture.
  Arms: Exposed d-PTFE

SUMMARY:
The aim of the current study is to compare the effect socket sealing with flowable resin composite compared to dense polytetrafluoroethylene membrane after filling the extraction site with xenograft particles in terms of soft and hard tissue changes, procedural time, post operative pain, patients' satisfaction, and cost effectiveness.

DETAILED DESCRIPTION:
Implant placement has become the gold standard for replacing missing teeth. One of the biggest challenges present when placing implants is the lack of sufficient bone dimensions. This deficiency may be a common finding due to the process of post extraction remodeling where both bone height and width are reduced, complicating implant placement. As a result, several procedures have been suggested to address this issue. Socket preservation is one of the most implemented procedures used today to limit the amount of bone lost during post extraction remodeling. The current study was designed to compare the effectiveness of using flowable composite resin for socket sealing as an alternative to using d-PTFE membranes, bypassing the added time, cost and trauma needed for tunnel preparation and membrane tucking.

ELIGIBILITY:
Inclusion Criteria:

* Patients having single non-adjacent hopeless maxillary tooth in the esthetic zone that are indicated for extraction.
* Patients with healthy systemic condition.
* Patients aged from 20 to 70 years old.
* Good oral hygiene.
* Accepts 4 months follow-up period (cooperative patients).

Exclusion Criteria:

* Systemic diseases or medications that might affect bone metabolism, increase surgical risk or complicate post-operative healing.
* Previous bone augmentation to implant site.
* Untreated periodontal diseases.
* Para-functional habits such as bruxism and clenching.
* History of radiation therapy to the head and neck.
* Heavy smokers (≥ 10 cigarettes per day).
* Pregnant or lactating females.
* Alcoholism or drug abuse.
* Psychiatric problems.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in horizontal bone dimension | 4 Months
  Cone beam computed tomography (CBCT) (Millimeters)

SECONDARY OUTCOMES:
Change in Vertical bone dimension | 4 Months
  Cone beam computed tomography (CBCT) (Millimeters)
Keratinized tissue thickness | 4 Months
  Millimeters
Procedural time | During surgery
  Stopwatch
Post-operative pain | 1 week
  Visual analogue scale (Santos, Botelho et al. 2021) (0-10) 0=No discomfort 10=Worst discomfort
Patient Satisfaction | 2 weeks
  Three questions questionnaire (Kiyak, Hohl et al. 1984). 7-point response scale:
  7= very likely (or very satisfied), 1= not at all likely (or not at all satisfied)
Incidence of complications | 4 Months
  Checklist

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of oral and dental medicine, Cairo university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided